CLINICAL TRIAL: NCT00948571
Title: Influence of Posture, Anesthesia and Surgical Technique on Airway Resistance of the Upper and Lower Airway and Lung Function.
Brief Title: Influence of Posture and Gas Insufflation on Perioperative Lung Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kliniken Essen-Mitte (Other)
Responsible Party: Prof. Dr. Harald Groeben, Kliniken Essen-Mitte
Other Study IDs: 06-3085
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Pneumoperitoneum
Keywords: Vital capacity, FEV1, airway resistance; perioperative changes in lung function
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- head down, laparoscopic: 20 patients with laparoscopic surgery (radical robotic prostatectomy) in head down position
- head down, open: 20 patients undergoing "open"surgery (open radical prostatectomy) in head down position.
- horizontal, open: 20 patients undergoing "open" surgery in horizontal position (open hemicolectomy)

SUMMARY:
Perioperative airway resistance and lung function are evaluated perioperatively in patients, who undergo surgical procedures in different postures and with or without gas insufflation into the peritoneal cavity.

DETAILED DESCRIPTION:
Lung function, upper and lower airway resistance measurements are performed in patients in prone horizontal or head tilted down (40°) position. Half of the patients with head down position will have surgery in laparoscopic technique (including gas insufflation to achieve a pneumoperitoneum). Measurements are performed on the day prior to surgery, on the morning of surgery, 30 - 45 minutes, 2 hours, and 24 hours after extubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age.
* Patients with normal lung function with respect to age, gender and weight. -Patients scheduled for Prostatectomies, robotic Prostatectomies, and open hemicolectomies.

Exclusion Criteria:

* Patients younger than 18 years.
* Patients with pathological lung function.
* Patients with with major cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients scheduled for "robotic" prostatectomies 20 patients scheduled for open prostatectomies 20 patients scheduled for open hemicolectomies
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-10 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of FEV1 (forced expiratory volume in one second) and the MEF50/MIF50 ratio | 18 months

SECONDARY OUTCOMES:
Changes in nasal airway resistance | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Harald Groeben, Prof. Dr., Principal Investigator — Klniken Essen-Mitte
Locations (1):
- Prof. Dr. Harald Groeben, Essen, Germany

REFERENCES:
- [Background] Craig DB. Postoperative recovery of pulmonary function. Anesth Analg. 1981 Jan;60(1):46-52. No abstract available. PMID 7006464
- [Background] Herbstreit F, Peters J, Eikermann M. Impaired upper airway integrity by residual neuromuscular blockade: increased airway collapsibility and blunted genioglossus muscle activity in response to negative pharyngeal pressure. Anesthesiology. 2009 Jun;110(6):1253-60. doi: 10.1097/ALN.0b013e31819faa71. PMID 19417617
- [Background] Chiu KL, Ryan CM, Shiota S, Ruttanaumpawan P, Arzt M, Haight JS, Chan CT, Floras JS, Bradley TD. Fluid shift by lower body positive pressure increases pharyngeal resistance in healthy subjects. Am J Respir Crit Care Med. 2006 Dec 15;174(12):1378-83. doi: 10.1164/rccm.200607-927OC. Epub 2006 Sep 22. PMID 16998093